CLINICAL TRIAL: NCT06370195
Title: Effect of Stellate Ganglion Block on Drooling in Parkinson's Syndrome: A Randomized Controlled Study
Brief Title: Effect of Stellate Ganglion Block on Drooling in Parkinson's Syndrome
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Babujinaya Cela (Other Government)
Responsible Party: Sponsor-Investigator, Babujinaya Cela, Research Director, Buraidah Central Hospital
Organization: Buraidah Central Hospital (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SGB-Liuxian
Record Dates: First submitted 2024-04-13; First posted 2024-04-17 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Parkinson's Syndrome
MeSH Terms: conditions — Parkinson Disease | interventions — Lidocaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Comprehensive rehabilitation+Stellate ganglion block (Experimental): Patients enrolled are firstly numbered for privacy with software and divided into the observation group and the control group with. Additionally, the staffs involved in assessment would not participate in the intervention of the study. The treatment lasts 10 days.
  Interventions: Behavioral: Comprehensive rehabilitation; Procedure: Stellate ganglion block; Drug: Lidocaine hydrochloride
- Comparator: Comprehensive rehabilitation+placebo (Placebo Comparator): Patients enrolled are firstly numbered for privacy with software and divided into the observation group and the control group with. Additionally, the staffs involved in assessment would not participate in the intervention of the study. The treatment lasts 10 days.
  Interventions: Behavioral: Comprehensive rehabilitation; Procedure: Placebo injection

INTERVENTIONS:
Behavioral: Comprehensive rehabilitation — The study lasted 10d for each patient. During the treatment, All the participants were provided with the rehabilitation therapy, which included routine rehabilitation, cognitive training, swallowing function training.
Procedure: Stellate ganglion block — Based on the invention above, the patients in the observation group were provided with Stellate ganglion block , using 1.5ml of 2% Lidocaine hydrochloride (1ml: 0.5mg) and 500ug of Vitamin B12 (1ml: 0.5g). The percutaneous approach via the paratracheal route was used for Stellate ganglion block . The operator stood on the side of the block, instructed the patient to lie supine with a thin pillow placed below the shoulders, and tilted the head 45° towards the blocked side, fully exposing the neck. Then, routine disinfection of the neck skin was performed. The puncture site was located 2.5 cm above the sternoclavicular joint and 1.5 cm lateral to the midline of the neck.
  Arms: Comprehensive rehabilitation+Stellate ganglion block
Drug: Lidocaine hydrochloride — Based on the invention above, the patients in the observation group were provided with Stellate ganglion block , using 1.5ml of 2% Lidocaine hydrochloride (1ml: 0.5mg) and 500ug of Vitamin B12 (1ml: 0.5g). The percutaneous approach via the paratracheal route was used for Stellate ganglion block . The operator stood on the side of the block, instructed the patient to lie supine with a thin pillow placed below the shoulders, and tilted the head 45° towards the blocked side, fully exposing the neck. Then, routine disinfection of the neck skin was performed. The puncture site was located 2.5 cm above the sternoclavicular joint and 1.5 cm lateral to the midline of the neck.
  Arms: Comprehensive rehabilitation+Stellate ganglion block
Procedure: Placebo injection — 1 milliliter of normal saline will be used for injection. The percutaneous approach via the paratracheal route was used for Stellate ganglion block . The operator stood on the side of the block, instructed the patient to lie supine with a thin pillow placed below the shoulders, and tilted the head 45° towards the blocked side, fully exposing the neck. Then, routine disinfection of the neck skin was performed. The puncture site was located 2.5 cm above the sternoclavicular joint and 1.5 cm lateral to the midline of the neck.
  Arms: Comparator: Comprehensive rehabilitation+placebo

SUMMARY:
This is a randomized controlled study, including dysphagic patients with Parkinson's syndrome who were received in the department of rehabilitation medicine. All patients are randomly allocated to the observation group or the control group. Both groups are provided with comprehensive rehabilitation. Besides, the observation group additionally undergoes the stellate ganglion block. At admission and after 10-day treatment, Functional Oral Intake Scale, Drooling amount, depression are assessed.

DETAILED DESCRIPTION:
Palliation of dysphagia in patients with Parkinson's syndrome continues to be a challenge.

This is a randomized controlled study, including dysphagic patients with Parkinson's syndrome who were received in the department of rehabilitation medicine. All patients are randomly allocated to the observation group or the control group. Both groups are provided with comprehensive rehabilitation. Besides, the observation group additionally undergoes the stellate ganglion block. At admission and after 10-day treatment, Functional Oral Intake Scale, Drooling amount, depression are assessed.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years.
* Meeting the diagnostic criteria for Parkinson's disease developed by the Neurology Branch of the Chinese Medical Association in 2006.
* Diagnosed with dysphagia confirmed by the video fluoroscopic swallowing study.
* Stable vital signs, conscious, able to cooperate with assessment and treatment.

Exclusion Criteria:

* Dysphagia possibly caused by other reasons, such as cerebrovascular disease, trauma, neuromuscular diseases, malignant diseases of the pharynx and larynx, and digestive tract diseases.
* History of mental diseases or use of antipsychotics.
* Complicated with cognitive impairment or consciousness dysfunction.
* Simultaneously suffering from severe liver, kidney failure, tumors, or hematological diseases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-04 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Drooling amount | day 1 and day 10
  All participants' saliva was collected within 5 minutes into a cup, followed by the comparison of saliva quantity, composition 1 hour before noon, the amount will be recorded.

SECONDARY OUTCOMES:
Modified Barthel Index | day 1 and day 10
  the activities of daily living of patients will be assessed using the modified Barthel Index . The scale includes 10 items such as feeding, bathing, walking, dressing. Each item is rated on a 4-point scale based on the level of assistance required, with a total score of 100 points. There is a positive correlation between activities of daily living and the final score.
Patient Health Questionnaire-9 | day 1 and day 10
  Patient Health Questionnaire-9 (PHQ-9) is a commonly used depression screening tool consisting of 9 items, designed to assess the severity of individual depressive symptoms. Each item is rated from 0 (not at all) to 3 (nearly every day) based on how the individual has been feeling over the past two weeks.
  The total score ranges from 0 to 27, and the severity of depressive symptoms is assessed as follows:
  0-4: Minimal depression 5-9: Mild depression 10-14: Moderate depression 15-19: Moderately severe depression 20 and above: Severe depression When assessing the severity of depressive symptoms, a higher total score indicates more severe symptoms, while a lower total score indicates milder symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Louis Wi, Study Director — Site Coordinator of United Medical Group